CLINICAL TRIAL: NCT07370649
Title: Long-Acting Cabotegravir And Rilipivirine In People Living With HIV-1 Subtype A6. A Multicentre Real-world, Retrospective Matched Case Study
Brief Title: Long-Acting Cabotegravir and Rilpivirine in People Living With HIV-1 Subtype A6: A Real-World Retrospective Study
Acronym: LACRIS
Status: Not yet recruiting | Type: Observational
Sponsor: Pomeranian Medical University Szczecin (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: LACRIS
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Human Immunodeficiency Virus (HIV)-1 Infection; HIV-1 Subtype A6 Infection; HIV-1 Subtype B Infection; Virologically Suppressed HIV-1 Infection Receiving Long-Acting Antiretroviral Therapy
Keywords: HIV-1; Long-Acting Antiretroviral Therapy; Cabotegravir; Rilpivirine; CAB/RPV LA; HIV-1 Subtype A6; HIV-1 Subtype B; Virologic Suppression; Real-World Study; Retrospective Study; Injectable HIV Therapy; Treatment Persistence; Virologic Failure
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — cabotegravir; Rilpivirine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Peripheral blood samples collected for routine clinical care, with proviral DNA extracted from blood cells for HIV-1 genotyping in participants with unknown subtype.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HIV-1 subtype A6: This cohort includes adults living with HIV-1 with a confirmed subtype A6 infection who received at least one dose of long-acting injectable cabotegravir plus rilpivirine (CAB/RPV LA) as part of routine clinical care. Participants are treatment-experienced and include individuals with suppressed or unsuppressed viral load at treatment initiation. Clinical outcomes, including virologic effectiveness, treatment persistence, adherence, and discontinuation, are assessed retrospectively using existing medical records. This cohort is matched with the subtype B cohort using propensity score methods.
  Interventions: Drug: Cabotegravir Plus Rilpivirine Long-Acting Injectable
- HIV-1 Subtype B Cohort: This cohort consists of adults living with HIV-1 with a confirmed subtype B infection who received long-acting injectable cabotegravir plus rilpivirine (CAB/RPV LA) in routine clinical practice. Participants are selected and matched to the subtype A6 cohort based on predefined confounding variables, including age, gender, body mass index category, and CD4 cell nadir. Outcomes are evaluated retrospectively to provide a comparative real-world context for the subtype A6 cohort.
  Interventions: Drug: Cabotegravir Plus Rilpivirine Long-Acting Injectable
- HIV-1 Subtype Unknown Cohort: This cohort includes adults living with HIV-1 who received long-acting injectable cabotegravir plus rilpivirine (CAB/RPV LA) and had no documented HIV-1 subtype at the time of treatment initiation. Participants are analyzed as an unmatched descriptive group. Retrospective clinical outcome data are collected from medical records. For selected participants, proviral DNA genotyping from blood samples is performed after initial analyses to explore the clinical relevance of HIV-1 subtype knowledge prior to switching to long-acting injectable therapy.
  Interventions: Drug: Cabotegravir Plus Rilpivirine Long-Acting Injectable

INTERVENTIONS:
Drug: Cabotegravir Plus Rilpivirine Long-Acting Injectable — Cabotegravir plus rilpivirine long-acting (CAB/RPV LA) is a complete antiretroviral regimen administered as intramuscular injections and approved for the maintenance treatment of HIV-1 infection in adults. In this observational, retrospective study, CAB/RPV LA is used as part of routine clinical care and is not assigned by the study protocol. Participants received CAB/RPV LA according to local prescribing information, including dosing intervals and injection windows.
  The study evaluates real-world clinical outcomes of CAB/RPV LA across different HIV-1 subtype groups (subtype A6, subtype B, and unknown subtype). Outcomes of interest include virologic effectiveness, treatment persistence, adherence to injection schedules, and treatment discontinuation. No study-specific modifications to dosing, administration, or clinical management are performed.
  Other Names: CAB/RPV LA; Long-Acting Cabotegravir and Rilpivirine; Cabotegravir + Rilpivirine

SUMMARY:
This study evaluates the real-world effectiveness and safety of a long-acting injectable HIV treatment consisting of cabotegravir and rilpivirine in people living with HIV-1. The focus is on individuals with HIV-1 subtype A6, which is common in Eastern Europe and among people who acquired HIV in that region, and on comparison with individuals with subtype B and those with an unknown subtype.

Although long-acting cabotegravir and rilpivirine are widely used and effective, limited real-world data are available on how well this treatment works in people with HIV-1 subtype A6. This is important because subtype A6 has been suggested as a potential risk factor for treatment failure, but current evidence is inconclusive.

The study uses existing medical records from treatment centers in Poland, Germany, and the Czech Republic. It includes adults with HIV who have received at least one injection of long-acting cabotegravir and rilpivirine and follows their clinical outcomes for up to 24 months. Researchers will assess viral suppression, treatment persistence, adherence to injection schedules, and reasons for treatment discontinuation.

The results of this study will help clinicians better understand whether HIV-1 subtype A6 affects treatment outcomes and whether knowing a patient's HIV subtype is important when deciding to switch to long-acting injectable therapy. The findings may support safer and more effective use of this treatment in diverse patient populations.

DETAILED DESCRIPTION:
This is a multicentre, international, real-world, retrospective observational study designed to evaluate clinical outcomes of long-acting injectable cabotegravir plus rilpivirine (CAB/RPV LA) in adults living with HIV-1. The study is conducted at HIV treatment centers in Poland, Germany, and the Czech Republic and is based on routinely collected clinical data from electronic medical records and paper charts.

The study population includes treatment-experienced individuals aged 18 years or older who received at least one dose of CAB/RPV LA in routine clinical practice. Participants are grouped according to HIV-1 subtype: subtype A6, subtype B, and unknown subtype. Individuals with known subtype A6 are matched with individuals with subtype B using propensity score matching to reduce the impact of confounding factors. Participants with unknown subtype are analyzed as an unmatched group.

Clinical data are collected from the time of CAB/RPV LA initiation (index date) and from follow-up visits closest to 6, 12, 18, and 24 months after initiation. Outcomes assessed include treatment persistence, adherence to injection schedules, discontinuation rates and reasons for discontinuation, and measures of virologic effectiveness. Virologic outcomes include viral suppression, viral rebound, and confirmed virologic failure as defined by standard HIV RNA criteria.

For participants with unknown HIV-1 subtype, proviral DNA genotyping is performed after initial descriptive analyses to explore whether knowledge of HIV-1 subtype has prognostic relevance for clinical outcomes. Genotypic data are analyzed descriptively and may inform additional exploratory analyses.

As this is a retrospective, non-interventional study using existing clinical data, no study-specific treatment interventions are performed. Safety data collection is limited to adverse events leading to treatment discontinuation, reflecting routine clinical practice. The study aims to provide clinically relevant real-world evidence on the use of CAB/RPV LA across different HIV-1 subtypes, with particular focus on subtype A6.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of HIV-1 infection
* Age ≥18 years at the time of initiation of long-acting cabotegravir plus rilpivirine (CAB/RPV LA)
* Received at least one dose of CAB/RPV LA as part of routine clinical care
* Availability of relevant clinical data in medical records for retrospective analysis
* Signed informed consent for use of clinical data
* Agreement to provide an additional blood sample for proviral DNA genotyping, if HIV-1 subtype was unknown at treatment initiation

Exclusion Criteria:

- Lack of patient consent for use of clinical data for research purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults aged 18 years or older living with HIV-1 infection who have received long-acting injectable cabotegravir plus rilpivirine (CAB/RPV LA) as part of routine clinical care. Participants are treatment-experienced and include individuals with suppressed or unsuppressed HIV-1 viral load at the time of treatment initiation.
  Patients are identified retrospectively from electronic medical records at participating HIV treatment centers in Poland, Germany, and the Czech Republic. Participants are grouped according to documented HIV-1 subtype (subtype A6, subtype B, or unknown subtype). Individuals with known subtype A6 are matched with individuals with subtype B based on selected clinical characteristics, while participants with unknown subtype are analyzed as an unmatched descriptive cohort.
  The study includes a broad, real-world patient population without upper age limits or sex-based restrictions, reflecting routine clinical practice in participating ce
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Virologic Suppression at Follow-Up | Up to 24 months after initiation of CAB/RPV LA
  Proportion of participants with HIV-1 RNA viral load <50 copies/mL at follow-up after initiation of long-acting cabotegravir plus rilpivirine (CAB/RPV LA), assessed using available clinical laboratory measurements. Virologic suppression will be evaluated at approximately 6, 12, 18, and 24 months after treatment initiation, with last observation carried forward where applicable.

SECONDARY OUTCOMES:
Treatment Persistence on CAB/RPV LA | Up to 24 months after initiation of CAB/RPV LA
  Proportion of participants who remain on long-acting cabotegravir plus rilpivirine (CAB/RPV LA) at each follow-up time point after initiation, based on documentation of continued injections in routine clinical care.
Treatment Discontinuation Rate | Up to 24 months after initiation of CAB/RPV LA
  Proportion of participants who discontinue CAB/RPV LA after initiation, including documentation of the reason for discontinuation such as adverse events, virologic failure, or other clinical or patient-related reasons.
Time to Treatment Discontinuation | Up to 24 months after initiation of CAB/RPV LA
  Median time from first administration of CAB/RPV LA to permanent discontinuation of the regimen, calculated using available clinical records.
Adherence to Injection Schedule | Up to 24 months after initiation of CAB/RPV LA
  Adherence to the CAB/RPV LA dosing schedule, assessed as the proportion of participants receiving injections within the allowed ±7-day dosing window relative to the target injection date.
Delayed or Missed Injections | Up to 24 months after initiation of CAB/RPV LA
  Proportion of participants with delayed injections (>7 days after target date), missed injections, and the number and duration of delayed or missed injections during follow-up.
Confirmed Virologic Failure (CVF) | Up to 24 months after initiation of CAB/RPV LA
  Proportion of participants meeting criteria for confirmed virologic failure, defined as two consecutive HIV-1 RNA measurements ≥200 copies/mL, or one HIV-1 RNA ≥200 copies/mL followed by treatment discontinuation within four months.
Viral Rebound | Up to 24 months after initiation of CAB/RPV LA
  Proportion of participants experiencing viral rebound, including viral blips (single HIV-1 RNA 50-199 copies/mL followed by <50 copies/mL), low-level viremia (two consecutive measurements 50-199 copies/mL), or viremia >200 copies/mL not leading to treatment discontinuation.
Virologic Non-Response After CVF | Up to 24 months after initiation of CAB/RPV LA
  Proportion of participants who do not achieve re-suppression (HIV-1 RNA <50 copies/mL) following confirmed virologic failure during the follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Katedra Chorób Zakaźnych i Niedoborów Immunologicznych, Szczecin, West Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this is a retrospective, observational study based on routinely collected clinical data from multiple centers. The data are pseudo-anonymized and subject to local data protection regulations and ethical approvals, which limit the ability to share individual-level data outside the study team.